CLINICAL TRIAL: NCT04977661
Title: A Randomized Study to Compare the Efficacy of Vitamin E, Ursodeoxycholic Acid and Pentoxyfylline on Egyptian Patients With Non-alcoholic Fatty Liver Disease Using (IL6 and CCL2) as a Predictors of Non-alcoholic Steatohepatitis
Brief Title: Comparing the Effects of Vitamin E, Ursodeoxycholic Acid and Pentoxyfylline on Egyptian Non-alcoholic Steatohepatitis (NASH) Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Aya Emad Nasr Mohammed Fouda, Dr assistant lecturer, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 154569224578
Record Dates: First submitted 2021-07-07; First posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Nonalcoholic Steatohepatitis (NASH)
Keywords: Vitamin E, Ursodeoxycholic acid, Pentoxifylline, NASH
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Vitamin E; alpha-Tocopherol; Ursodeoxycholic Acid; Pentoxifylline

STUDY DESIGN:
Intervention Model Description: prospective, randomized, and single blind study
Who Masked: Participant
Masking Description: (single blind study) : Participants did not know the treatment which was given
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group1 (Active Comparator): Group I (n = 34) received 400 IU Vitamin E (Vitamin E 400 IU®, MEPACO Pharmaceutical Company, Sharqia, Egypt) twice daily for 3 month
  Interventions: Drug: Vitamin E
- Group2 (Active Comparator): Group II (n =34) received 250 mg Ursodeoxycholic acid (Ursofalk 250 mg®, MINAPHARM Pharmaceutical Company, Cairo, Egypt) twice daily for 3 months
  Interventions: Drug: Ursodeoxycholic acid
- Group3 (Active Comparator): Group III (n = 34) received 400 mg sustained release (SR) Film-Coated Tablets of pentoxifylline (Trental 400 mg®, SANOFI Pharmaceutical Company, Cairo, Egypt) twice daily for 3 months
  Interventions: Drug: Pentoxifylline

INTERVENTIONS:
Drug: Vitamin E — Vitamin E is one of the body's most effective chain-breaking antioxidants that has shown to delay the pathogenesis of NASH.
  Other Names: Alpha-Tocopherol
  Arms: Group1
Drug: Ursodeoxycholic acid — is a metabolic by-product of intestinal bacteria and has been proven to be useful in the non-surgical treatment of cholesterol gallstones and primary biliary cirrhosis (PBC)
  Other Names: Ursofalk
  Arms: Group2
Drug: Pentoxifylline — it is a well-tolerated medication that improves blood
  viscosity and erythrocyte rheological characteristics in individuals with peripheral vascular disease 20. In addition, PTX is a nonspecific phosphodiesterase inhibitor that increases cyclic adenosine monophosphate (cAMP) levels while decreasing TNF-a gene transcription
  Other Names: Trental
  Arms: Group3

SUMMARY:
We conducted a 3-month, randomized, single-blind study in 102 Egyptian NASH patients who were divided into three groups; group 1 included 34 patients received Vit. E 400 mg twice a day, group 2 included 34 patients received UDCA 250 mg twice a day and group 3 included 34 patients received PTX 400 mg twice daily for 3 months. The following parameters were measured both before and after intervention intake; liver aminotransferases (AST, ALT), cytokine and chemokine (IL6 and CCL2/MPC-1), albumin, total bilirubin, direct bilirubin, total cholesterol, triglyceride, LDL, HDL.

DETAILED DESCRIPTION:
This was a 3-month, prospective, randomized, and single blind study. Participants were recruited from the outpatient clinic and hepatology, gastroenterology and infectious diseases department at Kafrelsheikh University Hospital between February 2020 and January 2021. Two-hundred and five Egyptian patients diagnosed with NAFLD with potential clinical inclusion criteria were invited for a screening session to determine their eligibility for the study. Patients were enrolled in the study if they are > 18 years old, had evidence for NASH; persistently elevated alanine aminotransferase (ALT) >1.5 times the upper limit of normal), imaging (ultrasound) showing fatty infiltration, and histological evidence of NASH after biopsy (macrovascular steatosis, ballooning degeneration of hepatocytes, scattered lobular inflammation and apoptotic bodies).One hundred and forty-six patients were excluded from the study either because they did not meet the inclusion criteria (n = 135) or refused to enroll in the study (n =11). Qualifying participants (n = 102) were randomly assigned to one of the three treatment groups using a computer-generated randomization sequence. Group I (n = 34) received 400 IU Vitamin E (Vitamin E 400 IU®, MEPACO Pharmaceutical Company, Sharqia, Egypt) twice daily for 3 months. Group II (n =34) received 250 mg Ursodeoxycholic acid (Ursofalk 250 mg®, MINAPHARM Pharmaceutical Company, Cairo, Egypt) twice daily for 3 months. Group III (n = 34) received 400 mg sustained release (SR) Film-Coated Tablets of pentoxifylline (Trental 400 mg®, SANOFI Pharmaceutical Company, Cairo, Egypt) twice daily for 3 months. Patients were followed up every week to ensure compliance, drug adherence and to report side effects or drop out from the study.The following parameters were measured both before and after intervention intake; liver aminotransferases (AST, ALT), cytokine and chemokine (IL6 and CCL2/MPC-1), albumin, total bilirubin, direct bilirubin, total cholesterol, triglyceride, LDL, HDL.

ELIGIBILITY:
Inclusion Criteria:

* Patients were enrolled in the study

  1. if they are > 18 years old
  2. had evidence for NASH; persistently elevated alanine aminotransferase (ALT) >1.5 times the upper limit of normal)
  3. imaging (ultrasound) showing fatty infiltration, and histological evidence of NASH after biopsy (macrovascular steatosis, ballooning degeneration of hepatocytes, scattered lobular inflammation and apoptotic bodies).

Exclusion Criteria:

* Patients were ruled out if they had

  1. history of alcohol dependence
  2. treatment with drugs known to induce NASH (e.g. amiodarone, calcium channel blocker, tamoxifen, oral anticoagulation, methotrexate , steroids and estrogen)
  3. positive serologic markers for known chronic liver diseases (hepatitis B surface antigen, anti-hepatitis C virus antibody antinuclear antibody)
  4. human immunodeficiency virus (HIV) infection
  5. Diabetes
  6. decompensated liver disease defined as serum bilirubin level >1 mg/dL, albumin level ˂3.5 g/dL, and international normalized ratio (INR) ≥1.7.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — > 18 years old
Enrollment: 102 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2021-01-10 (Actual)

PRIMARY OUTCOMES:
Resolution of NASH | 3 months
  Relieve clinical symptoms and prevent progression

SECONDARY OUTCOMES:
Normalization of hepatic aminotransferases(ALT and AST) | 3 months
  ALT and AST return to normal values

CONTACTS AND LOCATIONS:
Locations (1):
- Hepatology, gastroenterology and infectious diseases department at Kafrelsheikh University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available

REFERENCES:
- [Result] Younossi Z, Tacke F, Arrese M, Chander Sharma B, Mostafa I, Bugianesi E, Wai-Sun Wong V, Yilmaz Y, George J, Fan J, Vos MB. Global Perspectives on Nonalcoholic Fatty Liver Disease and Nonalcoholic Steatohepatitis. Hepatology. 2019 Jun;69(6):2672-2682. doi: 10.1002/hep.30251. PMID 30179269
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30179269/